CLINICAL TRIAL: NCT03759535
Title: Research on the Detection of Donor Derived Cell Free DNA （cfDNA）for the Early-stage Diagnosis of Acute Rejection Reaction Post Kidney Transplantation
Brief Title: Study in Detection cfDNA for the Early-stage Diagnosis of Acute Rejection Post-renal Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RenJiH-renal transplantation01
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-09

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: DNA acute rejection kidney transplantation
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Donor derived cell free DNA (dd-cfDNA) is utilized as a measure for "liquid biopsy", it is easy to operate, with less invasiveness, and it can reflect related conditions in a timely manner，etc.. This measure can detect the injury degree for allograft, and the index will rise before fluctuation reflection of the syndrome and related laboratory indexes, which is crucial for the very early-stage diagnosis of allograft acute rejection, and the further prevention of allograft injury. In the mean time, dd-cfDNA assumes high utilization value for the monitoring of immunosuppressive conditions, and therefore providing instructions for the optimization of the immunosuppressive treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control group and Case group: Control group:
  The allograft kidneys function normally. The rejection of allograft kidneys are excluded. The patients have no infectious complications.
  Case group:
  There is obvious evidence for acute rejection of the allograft kidneys. The patients have no infectious complications.
  Interventions: Diagnostic Test: Acute rejection

INTERVENTIONS:
Diagnostic Test: Acute rejection — Donor derived cell free DNA

SUMMARY:
Acute rejection (AR) is still one of the major complications after kidney transplantation. The current diagnosis measure for AR is primarily pathological puncture test and hematuria biomarker detection, yet due to their inferior performance on timeliness, the allograft kidneys usually have been in severe conditions when the diagnoses take place. Donor derived cell free DNA (dd-cfDNA) is utilized as a measure for "liquid biopsy", it can predict acute rejection at very early periods, and it is easy to operate, with fewer invasive injuries, and can reflect related conditions in a timely manner, etc.. This study plans to utilize second-generation sequencing technology to systematically evaluate the abundance variations of nuclear genome and mitocondria derived dd-cfDNA in the kidney transplant recipients' blood and urine, thus it can assist in accumulating more proof for the clinical utilization of dd-cfDNA from different sources at the early stages of AR in evidence-based medicine, and lay foundation for the development of dd-cfDNA based early-stage rejection detection tools afterkidney transplantation surgery.

DETAILED DESCRIPTION:
With the growing development of kidney transplant technologies and immunosuppressive therapies, the number of end-stage renal disease patients receiving kidney transplant has been increasing. Acute rejection (AR) is one of the main complications for kidney transplantation, and AR is the major reason for lowering graft survival rate and for graft malfunction, thus the timely detection of AR and early interventions are crucial. The current clinical measures for the detection of AR include pathological puncture test and hematuria biomarker detection. Yet pathological tests are invasive, limited to sampling errors and the existing perception differences among observants, and with other disadvantages such as expensiveness, poor patient compliance, and related complications. Hematuria biomarker detection is slow in response and low in the sensitivity and specificity for reflecting the organs' metabolic index in the diagnosis of acute rejection injury. Though the monitoring of immunosuppressant drugs, immune molecules and cytokines in the blood circulation can both provide certain value for the evaluation of patients' immune status after organ transplant, these factors are not good indicators for the early-stage diagnosis of allograft injury. Donor derived cell free DNA (dd-cfDNA) is utilized as a measure for "liquid biopsy", it is easy to operate, with less invasiveness, and it can reflect related conditions in a timely manner, etc.. This measure can detect the injury degree for allograft, and the index will rise before fluctuation reflection of the syndrome and related laboratory indexes, which is crucial for the very early-stage diagnosis of allograft acute rejection, and the further prevention of allograft injury. In the mean time, dd-cfDNA assumes high utilization value for the monitoring of immunosuppressive conditions, and therefore providing instructions for the optimization of the immunosuppressive treatment.

Under the condition of signed informed consent, the study protocols were scheduled as below:

Self-control study protocol:

20 to-receive-kidney-transplant patients are randomized, the self-control study protocol is utilized for each patient as the following.

Before the kidney transplant surgery, 1ml of peripheral EDTA anticoagulant from the recipients, and 1ml of peripheral EDTA anticoagulant from the donors are collected.

In 1 week, 2 weeks, 3 weeks' time after the kidney transplant surgeries, 8 to 10 ml of peripheral blood from the recipients using cfDNA blood collection tubes, and 10 to 15 ml of midstream urine are collected respectively.

Inclusion criteria:

*Patients are suitable for kidney transplant surgeries.

Exclusion criteria:

* Patients have failed in the transplant surgeries.
* Patients have no urine 1 week after the transplant surgeries.
* Patients have severe infectious complications after the transplant surgeries. b, Case group: For 20 patients that have been diagnosed with acute rejection on the first visits, 8 to 10 ml of EDTA anticoagulant, 10 to 15 ml of midstream urine, 5 ml of saliva are collected before the treatment, 1 week and 2 weeks after the adjustment of the anti-rejection treatment, 8 to 10 ml of blood using cfDNA blood collection tubes, 10 to 15 ml of midstream urine, 5 ml of saliva are collected respectively.

Inclusion criteria:

Control group:

* The allograft kidneys function normally.
* The rejection of allograft kidneys are excluded.
* The patients have no infectious complications.

Case group:

* There is obvious evidence for acute rejection of the allograft kidneys.
* The patients have no infectious complications.

Exclusion criteria:

* The patients have infectious complications.
* The patients have tumors.
* The patients are pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Patients are suitable for kidney transplant surgeries. Or There is obvious evidence for acute rejection of the allograft kidneys. The patients have no infectious complications.

Exclusion Criteria:

* Patients have failed in the transplant surgeries. Patients have no urine 1 week after the transplant surgeries. Patients have severe infectious complications after the transplant surgeries. Or:The patients have infectious complications. The patients have tumors. The patients are pregnant.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 20 to-receive-kidney-transplant patients are randomized, the self-control study protocol is utilized for each patient as the following.
  Under the condition of signed informed consent, for 20 kidney transplant recipients For 20 patients that have been diagnosed with acute rejection on the first visits.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Renal allograft injury Renal allograft injury | 2 months
  serum creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Ming, Doctor, Study Director — RenJi Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] De Vlaminck I, Martin L, Kertesz M, Patel K, Kowarsky M, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Nicolls MR, Cornfield D, Weill D, Valantine H, Khush KK, Quake SR. Noninvasive monitoring of infection and rejection after lung transplantation. Proc Natl Acad Sci U S A. 2015 Oct 27;112(43):13336-41. doi: 10.1073/pnas.1517494112. Epub 2015 Oct 12. PMID 26460048
- [Result] Lo YM, Tein MS, Pang CC, Yeung CK, Tong KL, Hjelm NM. Presence of donor-specific DNA in plasma of kidney and liver-transplant recipients. Lancet. 1998 May 2;351(9112):1329-30. doi: 10.1016/s0140-6736(05)79055-3. No abstract available. PMID 9643800